CLINICAL TRIAL: NCT03980184
Title: The Use of Guanfacine (GUA) (3mg/Day) to Reduce Drug Craving, Improve Cognitive Flexibility and Result in Associated Lower Drug Use in Women With Substance Use Disorder (SUD).
Brief Title: Guanfacine to Improve Substance Use Outcomes in Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, RAJITA SINHA, Professor, Department of Psychiatry,, Yale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2000023100; 1R01DA047094-01A1 (NIH)
Record Dates: First submitted 2019-03-29; First posted 2019-06-10 (Actual); Results first posted 2024-01-08 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Guanfacine; Behavior Therapy

STUDY DESIGN:
Intervention Model Description: randomized double blind, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Study Medication (Experimental): guanfacine 3mg/day (GUA)
  Interventions: Drug: Guanfacine; Other: Behavioral Counseling
- placebo (Placebo Comparator): placebo (PBO)
  Interventions: Drug: Guanfacine; Other: Behavioral Counseling

INTERVENTIONS:
Drug: Guanfacine — Guanfacine 3mg/day Versus Placebo
  Other Names: Tenex,
Other: Behavioral Counseling — placebo
  Other Names: Manualized Drug Counseling

SUMMARY:
Hypothesis: Guanfacine (GUA) (3mg/day) will reduce drug craving, improve cognitive flexibility and result in associated lower drug use in women with substance use disorder (SUD) in an outpatient clinical setting.

DETAILED DESCRIPTION:
This study proposes to extend previous Phase I experimental work to address the following specific aims: (1) assess GUA's target engagement of drug craving and cognitive flexibility in a laboratory challenge session and in a 10-week outpatient clinical study, (2) demonstrate target validation by showing that reduced drug craving and improved cognitive flexibility will predict lower drug use outcomes during the 10-week clinical trial in SUD women, and finally, (3) evaluate data replication and scalability of GUA target effects across two clinical sites (Yale and SUNY-Stony Brook).

ELIGIBILITY:
Inclusion Criteria:

* 100 treatment seeking women
* Ages 18-70 years
* Body mass index (BMI) of 18-35
* Meet current DSM-V criteria for co-occurring SUDs, with primary DSM-V cocaine or primary DSM-V opioid use disorder AND co-occurring cannabis or alcohol or nicotine use disorders;
* Positive drug urine toxicology screens for primary addictive disorder during a 2-week intake assessment period
* Good health as verified by screening examination
* Able to read English and complete study evaluations
* Able to provide informed written and verbal consent

Exclusion Criteria:

* Meet criteria for physiological dependence on alcohol requiring medical detoxification
* Regular use of anti-hypertensives, anti-arrythmics, antiretroviral medications, and medications that would interact with Guanfacine and be contraindicated as per study physician;
* Psychotic or otherwise severely psychiatrically disabled (i.e., suicidal, homicidal, current mania)
* Significant underlying medical conditions which in the opinion of study physician would preclude patient from fully cooperating or be of potential harm during the course of the study; Specifically hepatic and renal impairment as per liver enzymes at 3X the normal limit, or BUN>50mg or BUN:Cr > 10:1.
* Hypotensive women with sitting blood pressure below 100/50 mmHG
* Women who are pregnant, nursing or refuse to use a reliable form of birth control
* EKG evidence at baseline screening of any clinically significant conduction abnormalities, including a Bazlett's QT c>470 msec for women.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — treatment seeking women
Enrollment: 74 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajita Sinha, PhD, Principal Investigator — Yale University
Locations (1):
- The Yale Stress Center: Yale University, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Medication | Placebo
Started (Participants randomized) | 38 | 36
Began Treatment | 36 | 34
Completed | 25 | 21
Not Completed | 13 | 15
Not completed — Dropped out before treatment | 2 | 2
Not completed — Lost to Follow-up | 11 | 13

BASELINE CHARACTERISTICS:
Population: Data represented here is from participants that started treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Medication | Placebo | Total
Number analyzed (Participants) | 36 | 34 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (12.5) | 40.1 (12.5) | 40 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 34 | 70
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — These are presented as individual rows because the categories are not exclusive (participants could identify with more than 1 category).
  Participants
    Caucasian | 20 | 23 | 43
    Black | 10 | 9 | 19
    Other | 6 | 2 | 8
    Hispanic | 7 | 3 | 10
Region of Enrollment [Number; unit: participants]
  United States | 36 | 34 | 70
Education [Mean (Standard Deviation); unit: years] | 13.4 (2.1) | 13.2 (2) | 13.3 (2.1)
Married/Cohabitating [Count of Participants; unit: Participants] | 6 | 6 | 12
Number of participants that used cocaine in the past 30 days [Count of Participants; unit: Participants] | 26 | 26 | 52
Mean days cocaine use in the past 30 days [Mean (Standard Deviation); unit: days] | 14 (12.1) | 11.0 (8.7) | 12.7 (10.6)
Number of participants that used opioids in the past 30 days [Count of Participants; unit: Participants] | 25 | 23 | 48
Mean days opioid use in the past 30 days [Mean (Standard Deviation); unit: days] | 12.1 (12.7) | 20.6 (11.5) | 16.4 (12.6)
Number of participants that used cannabis in the past 30 days [Count of Participants; unit: Participants] | 27 | 24 | 51
Mean days cannabis use in the past 30 days [Mean (Standard Deviation); unit: days] | 19.7 (11.3) | 20 (12.7) | 19.8 (11.8)
Number of participants that used alcohol in the past 30 days [Count of Participants; unit: Participants] | 31 | 30 | 61
Mean days alcohol use in the past 30 days [Mean (Standard Deviation); unit: days] | 15 (10.1) | 13.8 (8.9) | 14.4 (9.5)
Number of participants that used tobacco in the past 30 days [Count of Participants; unit: Participants] | 30 | 31 | 61
Mean days tobacco use in the past 30 days [Mean (Standard Deviation); unit: days] | 28.1 (6) | 29.2 (4.5) | 28.7 (5.3)
Addiction Severity Index Score (ASI) [Mean (Standard Deviation); unit: score on a scale] — 12 items with total score range 0-12 with higher scores indicating higher severity of addiction
  score on a scale | 6.6 (2.5) | 6.4 (2.5) | 6.5 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Drug Use With Substance Use Calendar
Description: Days of any drug use during the 10 week period (assessed daily and weekly via self report). Data presented here is the average between week 10 and week 1.
Time Frame: 10 weeks
Population: Participants who were randomized and received treatment.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Study Medication | Placebo
Number analyzed (Participants) | 36 | 34
days | -6.35 (1) | -5.61 (0.96)
Statistical Analysis 1: Comparison: Study Medication vs Placebo; Test type: Superiority; p = 0.08, Fisher Exact

2. Primary Outcome: Change in Abstinence Days
Description: Substance use calendar self report of daily drug use during 10 week treatment periods. Data presented here is the average between week 10 and week 1.
Time Frame: 10 weeks
Population: Participants who were randomized and received treatment.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Study Medication | Placebo
Number analyzed (Participants) | 36 | 34
days | 0.28 (0.25) | -0.12 (0.24)
Statistical Analysis 1: Comparison: Study Medication vs Placebo; Test type: Superiority; p < .001, Fisher Exact

3. Secondary Outcome: Change in Average Drug Craving
Description: Sum of average drug craving measured using Craving Questionnaires for cocaine, opiates, alcohol, nicotine and cannabis.The possible range for the average craving measure is 0 - 100. A higher score on the measure = greater avg drug craving.
Time Frame: 10 weeks
Population: Participants who were randomized and received treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Medication | Placebo
Number analyzed (Participants) | 36 | 34
score on a scale | -14.6 (4.4) | -21.9 (5.9)
Statistical Analysis 1: Comparison: Study Medication vs Placebo; Test type: Superiority; p = 0.703, Fisher Exact

4. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Event
Description: The Systematic Assessment of Treatment Emergent Events (SAFTEE) Questionnaire will be used to assess adverse events weekly during the trial. Data presented here is the number of participants that had any adverse events while on study.
Time Frame: 10 weeks
Population: Participants who were randomized and received treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Medication | Placebo
Number analyzed (Participants) | 36 | 34
Participants | 21 | 15

5. Other Pre Specified Outcome: Change in Stress Scores
Description: Repeated assessment of 14-item Perceived Stress Scale (score range: 0-53, higher scores are worse) assessed weekly. Scores are the average change between week 10 and week 1.
Time Frame: 10 weeks
Population: Participants who were randomized and received treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Medication | Placebo
Number analyzed (Participants) | 36 | 34
score on a scale | -2.8 (2.9) | 7.8 (2.8)
Statistical Analysis 1: Comparison: Study Medication vs Placebo; Test type: Superiority; p = 0.002, Fisher Exact

6. Other Pre Specified Outcome: Change in Anxiety Levels
Description: Repeated assessment of 14-item Hamilton Anxiety Scale (score range: 0-56, higher score is worse outcome) assessed weekly over 10 weeks. Scores are the average change between week 10 and week 1.
Time Frame: 10 weeks
Population: Participants who were randomized and received treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Medication | Placebo
Number analyzed (Participants) | 36 | 34
score on a scale | -1.9 (2.2) | -0.8 (1.3)
Statistical Analysis 1: Comparison: Study Medication vs Placebo; Test type: Superiority; p = 0.647, Fisher Exact

7. Other Pre Specified Outcome: Change in Depression Levels
Description: Repeated assessment of 17-item Hamilton Depression Scale (score range: 0-53, higher score is worse outcome) assessed weekly over 10 weeks. Scores are the average change between week 10 and week 1.
Time Frame: 10 weeks
Population: Participants who were randomized and received treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Medication | Placebo
Number analyzed (Participants) | 36 | 34
score on a scale | 0.5 (2.3) | 0.6 (1.4)
Statistical Analysis 1: Comparison: Study Medication vs Placebo; Test type: Superiority; p = 0.887, Fisher Exact

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Study Medication | Placebo
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/36
Serious Adverse Events (participants affected / at risk) | 2/36 | 4/34
Other Adverse Events (participants affected / at risk) | 19/36 | 11/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Medication (N=36) | Placebo (N=34)
General disorders and administration site conditions - Other, specify (General disorders) | 1 | 0 — Due to preexisting seizure condition
General disorders and administration site conditions - Other, specify (General disorders) | 1 | 0 — Wound treatment after stabbing
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 1 — Blood clot in leg and swelling
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 | 1 — Subject jumped from 3rd story window
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 1 — Admission due to zanax & ketamine misuse
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 1 — Inpatient drug rehab
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Medication (N=36) | Placebo (N=34)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Asthma
Dizziness (Nervous system disorders) | 4 | 1
Somnolence (Nervous system disorders) | 1 | 1 — Drowsiness
Dry mouth (Gastrointestinal disorders) | 8 | 0
Fever (General disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 2
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 1 — Head Feels Warm
Nervous system disorders - Other, specify (Nervous system disorders) | 2 | 0 — Numbness
General disorders and administration site conditions - Other, specify (General disorders) | 2 | 0 — Nosebleed
Pain (General disorders) | 4 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 — Itching
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 6 | 3 — Nausea/vomiting
Diarrhea (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 2 | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0 — Lessened Appetite
Fatigue (General disorders) | 3 | 3
General disorders and administration site conditions - Other, specify (General disorders) | 2 | 3 — Swelling
General disorders and administration site conditions - Other, specify (General disorders) | 1 | 0 — Sweatiness/Shakes
General disorders and administration site conditions - Other, specify (General disorders) | 2 | 1 — Tingling Sensation
Irregular menstruation (Reproductive system and breast disorders) | 2 | 0 — Change in Menstruation
Vascular disorders - Other, specify (Vascular disorders) | 3 | 1 — Hot and cold flashes
Vascular disorders - Other, specify (Vascular disorders) | 0 | 1 — Elevated Blood Pressure
Vascular disorders - Other, specify (Vascular disorders) | 1 | 0 — Decreased Blood Pressure
Psychiatric disorders - Other, specify (Psychiatric disorders) | 2 | 0 — Panic Attack
Tinnitus (Ear and labyrinth disorders) | 0 | 1
General disorders and administration site conditions - Other, specify (General disorders) | 2 | 0 — Sleep Problems

LIMITATIONS AND CAVEATS:
Small sample sizes, sample being limited to men were limitations. Caveats include small sample size limited examining treatment effects for specific drug use. Also, medication compliance moderated guanfacine effects on primary and secondary outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-10): https://cdn.clinicaltrials.gov/large-docs/84/NCT03980184/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-10): https://cdn.clinicaltrials.gov/large-docs/84/NCT03980184/ICF_001.pdf